CLINICAL TRIAL: NCT06153693
Title: A Randomized, Double-Blind, Placebo Controlled, Parallel Arm, Multicenter Phase 3 Study to Evaluate the Efficacy and Safety of Lorundrostat in Subjects With Uncontrolled and Resistant Hypertension
Brief Title: Efficacy and Safety of Lorundrostat in Subjects With Uncontrolled and Resistant Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mineralys Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MLS-101-301
Record Dates: First submitted 2023-11-17; First posted 2023-12-01 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Hypertension
Keywords: Blood pressure; Hypertension; Hypertensive; Resistant hypertension; Uncontrolled hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo once daily (QD) for 12 weeks
  Interventions: Drug: Placebo
- Dose 1 (Experimental): 50 mg lorundrostat Dose 1 once daily (QD) for 12 weeks
  Interventions: Drug: lorundrostat Dose 1
- Dose 2 (Experimental): 50 mg lorundrostat Dose 1 once daily (QD) for 6 weeks then 100 mg lorundrostat Dose 2 once daily (QD) for 6 weeks for subjects who meet prespecified criteria
  Interventions: Drug: lorundrostat Dose 2

INTERVENTIONS:
Drug: Placebo — Placebo once daily (QD) for 12 weeks
  Arms: Placebo
Drug: lorundrostat Dose 1 — 50 mg lorundrostat Dose 1 once daily (QD) for 12 weeks
  Arms: Dose 1
Drug: lorundrostat Dose 2 — 50 mg lorundrostat Dose 1 once daily (QD) for 6 weeks then 100 mg lorundrostat Dose 2 once daily (QD) for 6 weeks for subjects who meet prespecified criteria
  Arms: Dose 2

SUMMARY:
This is a Phase 3 trial to evaluate the BP-lowering effect of lorundrostat (an aldosterone synthase inhibitor) in subjects with uncontrolled and resistant hypertension taking between 2 and 5 anti-hypertensive (AHT) medications.

DETAILED DESCRIPTION:
This study is a Phase 3 trial to evaluate the BP-lowering effect of lorundrostat (an aldosterone synthase inhibitor) in subjects with uncontrolled and resistant hypertension taking between 2 and 5 anti-hypertensive (AHT) medications, one of which must be a thiazide or thiazide-like diuretic.

The study consists of a 2-week screening period with a 2-week single-blind run-in period followed by a 12-week randomized, double-blind, placebo-controlled, parallel arm period. Following the randomized period subjects will be offered an opportunity to participate in an open-label extension (OLE) study. Any subject electing to not participate in the OLE will undergo an end of study (EoS) visit, which will occur after end of treatment (EoT), to complete their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age at the time of signing the informed consent form (ICF)
2. At Screening and Randomization: AOBP SBP of ≥135 and ≤180 mmHg plus AOBP DBP of ≥65 and ≤110 mmHg, or AOBP DBP of ≥90 and ≤110 mmHg
3. Taking between 2 and 5 AHT medications,
4. History of hypertension lasting at least 6 months prior to Screening
5. Body mass index (BMI) of ≥18 kg/m2 at Screening

Exclusion Criteria:

1. Women who are pregnant, plan to become pregnant, or are breastfeeding
2. Participation in a study involving any investigational device or small-molecule drug within 4 weeks or 6 months for biologic (antibody) drugs prior to the Screening Visit
3. eGFR <45 mL/min/1.73m2 at Screening, calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula
4. Serum potassium >5.0 mmol/L at Screening or >4.8 mmol/L at Randomization
5. Serum sodium <135 mmol/L (corrected for hyperglycemia) at Screening.
6. History of heart failure, myocardial infarction, stroke, or transient ischemic attack within 6 months prior to the Screening Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1083 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Change from baseline in automated office BP (AOBP) SBP at Week 6 in subjects randomized to lorundrostat 50 mg QD compared to subjects randomized to placebo | Week 6

SECONDARY OUTCOMES:
Proportion of subjects with AOBP SBP <130 mmHg at Week 6 in subjects randomized to lorundrostat 50 mg QD compared to subjects randomized to placebo | Week 6
Change from baseline in AOBP SBP at Week 12 in subjects randomized to lorundrostat 50 mg QD with escalation to lorundrostat 100 mg QD compared to subjects randomized to placebo | Week 12
Change from baseline in AOBP SBP at Week 6 in subjects with uncontrolled hypertension on 2 prescribed AHT medications | Week 6
  Change from baseline in AOBP SBP at Week 6 in subjects with uncontrolled hypertension on 2 prescribed AHT medications randomized to lorundrostat 50 mg QD compared to subjects with uncontrolled hypertension on 2 prescribed AHT medications randomized to placebo
Change from baseline in AOBP SBP at Week 6 in subjects with uncontrolled hypertension on 3 or more prescribed AHT medications | Week 6
  Change from baseline in AOBP SBP at Week 6 in subjects with uncontrolled hypertension on 3 or more prescribed AHT medications (resistant hypertension) randomized to lorundrostat 50 mg QD compared to subjects with uncontrolled hypertension on 3 or more prescribed AHT medications (resistant hypertension) randomized to placebo
Change from baseline in AOBP SBP at Week 6 by obesity status in subjects randomized to lorundrostat 50 mg QD compared to subjects randomized to placebo | Week 6
Change from baseline in AOBP SBP at Week 12 in subjects who were escalated to lorundrostat 100 mg QD at week 6 (within-subjects analysis) | Week 12

CONTACTS AND LOCATIONS:
Locations (184):
- United States (87):
  - Advanced Cardiovascular, LLC - Alexander City Office, Alexander City, Alabama
  - Central Research Associates, Inc, Birmingham, Alabama
  - Cardiology, P.C., Birmingham, Alabama
  - Synexus (Radiant Research, Inc) - Alabama - Simon Williamson Clinic Location, Birmingham, Alabama
  - G & L Research LLC - Foley, Foley, Alabama
  - Accel Research Sites (ARS) - Birmingham Clinical Research Unit, Vestavia Hills, Alabama
  - Del Sol Research, Tucson, Arizona
  - Entertainment Medical Group, Inc., Beverly Hills, California
  - Amicis Research Center - Granada Hills, Granada Hills, California
  - Amicis Research Center - Northridge, Granada Hills, California
  - Marvel Clinical Research, LLC, Huntington Beach, California
  - Amicis Research Center, Northridge, California
  - Pasadena Clinical Trials, Pasadena, California
  - Empire Clinical Research (ECR), Pomona, California
  - Clinical Trials Research (CTR) - Sacramento, Sacramento, California
  - North America Research Institute, San Dimas, California
  - Amicis Research Center - Valencia, Valencia, California
  - CMR of Greater New Haven, Hamden, Connecticut
  - Chase Medical Research, LLC - Hamden, Waterbury, Connecticut
  - Indago Research and Health Center, Hialeah, Florida
  - Clinical Neuroscience Solutions (CNS Healthcare) - Jacksonville, Jacksonville, Florida
  - Nuovida Research Center Corp, Miami, Florida
  - Clinical Neuroscience Solutions (CNS Healthcare) - Orlando Research Center, Orlando, Florida
  - AES Orlando, Orlando, Florida
  - Patron Medical - Andres Patron D.O. (Patron Ventures, LLC), Pembroke Pines, Florida
  - Pines Care Research Center, LLC, Pembroke Pines, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Clinical Research of West Florida (CRWF) - Clearwater, Tampa, Florida
  - AES The Villages, The Villages, Florida
  - Morehouse School of Medicine (MSM), Atlanta, Georgia
  - ClinCept, LLC, Columbus, Georgia
  - Accel Research Sites- Decatur, Decatur, Georgia
  - Georgia Clinical Research Center, Inc, Lawrenceville, Georgia
  - Elite Clinical Trials, Blackfoot, Idaho
  - Rocky Mountain Diabetes Center, Idaho Falls, Idaho
  - Solaris Clinical Research (SCR), Meridian, Idaho
  - Synexus (Radiant Research, Inc) - Chicago, Chicago, Illinois
  - Healthcare Research Network-Chicago, Illinois (Flossmoor) Location, Flossmoor, Illinois
  - Koch Family Medicine, S.C., Morton, Illinois
  - Southern Illinois University School of Medicine - SIU Clinics - SIU Internal Medicine, Springfield, Illinois
  - Investigators Research Group LLC, Brownsburg, Indiana
  - Franciscan Physician Network, Indianapolis, Indiana
  - ASHA Clinical Research- Munster, LLC, Munster, Indiana
  - Synexus (Radiant Research, Inc) - Evansville, Newburgh, Indiana
  - Louisville Metabolic and Atherosclerosis Research Center (L-MARC), Louisville, Kentucky
  - Tulane Doctors - Heart & Vascular - Metairie, New Orleans, Louisiana
  - The Alliance for Multispecialty Research LLC (AMR) - Louisiana, New Orleans, Louisiana
  - Northwest Louisiana Nephrology, LLC - Shreveport, Shreveport, Louisiana
  - Grace Research, LLC, Shreveport, Louisiana
  - Boston Clinical Trials (BCT), Boston, Massachusetts
  - ActivMed Practices and Research, Methuen, Massachusetts
  - Hattiesburg Clinic - Medisync Clinical Research, Petal, Mississippi
  - Healthcare Research Network-Hazelwood, Hazelwood, Missouri
  - Clinical Research Consultants (CRC) - Kansas City, Kansas City, Missouri
  - Quality Clinical Research Inc. (QCR) - Omaha, Omaha, Nebraska
  - Synexus (Radiant Research, Inc) - Nevada - Rita B. Chuang, MD, Henderson, Nevada
  - Sierra Clinical Research-Las Vegas, Las Vegas, Nevada
  - Renown Regional Medical Center (Washoe Medical Center), Reno, Nevada
  - Synexus (Radiant Research, Inc) - New York, Jamaica, New York
  - North Shore Diabetes and Endocrine Associates (NSDEA) - New Hyde Park, New Hyde Park, New York
  - Columbia University, New York, New York
  - Randolph Health Internal Medicine/ Triad Internal Medicine, Asheboro, North Carolina
  - East Carolina University (ECU) Physicians - East Carolina Heart Institute - East Carolina University Location, Greenville, North Carolina
  - Physicians East, P.A. - Endocrinology, Greenville, North Carolina
  - Carteret Medical Group - Morehead City, Morehead City, North Carolina
  - Lucas Research, Inc. (Diabetes & Endocrinology Consultants PC) (DEC), New Bern, North Carolina
  - Diabetes & Endocrinology Associates of Stark County, Canton, Ohio
  - Lynn Institute of Norman (LION Research), Norman, Oklahoma
  - Valley Kidney Specialists PC - Allentown Cedar Crest, Bethlehem, Pennsylvania
  - Preferred Primary Care Physicians - Pleasant Hills - Curry Hollow Rd Location, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians (PPCP) - Uniontown - Jacob Murphy Lane Location, Uniontown, Pennsylvania
  - Chattanooga Medical Research (CMR), LLC, Chattanooga, Tennessee
  - The Alliance for Multispecialty Research LLC (AMR) - Knoxville (Volunteer Research Group), Knoxville, Tennessee
  - Clinical Neuroscience Solutions, Inc, Memphis, Tennessee
  - Punzi Medical Center and Trinity Hypertension Research Institute, Carrollton, Texas
  - AES Dallas Fort Worth, Dallas, Texas
  - Synergy Groups Medical, Houston, Texas
  - Juno Research, LLC, Houston, Texas
  - Discovery Clinical Trials (DCT) - McAllen, McAllen, Texas
  - Synergy Groups Medical - Missouri City, Missouri City, Texas
  - North Texas Family Medicine (NTFM) - Plano Office, Plano, Texas
  - Sun Research Institute (SRI) - San Antonio, San Antonio, Texas
  - Discovery Clinical Trials (DCT) - San Antonio, San Antonio, Texas
  - Global AES - Salt Lake City, Salt Lake City, Utah
  - Velocity Clinical Research - Salt Lake City (Advanced Clinical Research), West Jordan, Utah
  - Burke Internal Medicine, Burke, Virginia
  - Eastern VA Medical School, Norfolk, Virginia
- Australia (12):
  - Castle Hill Medical Centre, Castle Hill, New South Wales
  - Renal Research - Gosford, Gosford, New South Wales
  - University of Newcastle - John Hunter Hospital (JHH), Waratah, New South Wales
  - University of the Sunshine Coast - Clinical Trials Centre, Sippy Downs, Queensland
  - South Coast Renal, Southport, Queensland
  - AusTrials - Taringa, Taringa, Queensland
  - AusTrials - Wellers Hill, Taringa, Queensland
  - Fusion Clinical Research, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Dobney Hypertension Centre/ Royal Perth Hospital, Perth, Western Australia
  - Austin Health - Heidelberg Repatriation Hospital, Heidelberg Heights
  - AusTrials - Sunshine, St Albans
- Bulgaria (6):
  - Medical Center New Polyclinic Gabrovo Ltd., Gabrovo
  - Medical center Exacta Medica, Pleven
  - Medical Center Hera EOOD - Sofia, Sofia
  - ASOMHIDC (Ambulatory of specialized outpatient medical help in internal diseases and cardiology), Sofia
  - Medical Centre Zara-Med, Stara Zagora
  - DCC 1 - Veliko Tarnovo, Veliko Tarnovo
- Canada (3):
  - University of Alberta, Edmonton, Alberta
  - Stephen S. Chow Medicine Professional Corporation, East York, Ontario
  - Centre Medical L'Acadie - Montreal, Montreal, Quebec
- France (5):
  - Centre Hospitalier Annecy Genevois (CHANGE) - Site d'Annecy -, Annecy
  - Centre Hospitalier Universitaire (CHU) de Bordeaux - Hospitalier Saint-Andre, Bordeaux
  - Centre Hospitalier Universitaire de Nimes (CHU) - Hopital Universitaire Caremeau, Nîmes
  - Centre Hospitalier Universitaire (CHU) de Saint-Etienne - Hopital Nord, Saint-Priest-en-Jarez
  - Hopitaux Universitaires de Strasbourg - Le Nouvel Hopital Civil (NHC), Strasbourg
- Germany (10):
  - kfgn Site Operations & Services GmbH (KFGN) - Klinische Forschung Hannover-Mitte GmbH (KFHM), Hanover, Lower Saxony
  - Pfuetzner Science & Health Institute GmbH (PSHI) - Diabeteszentrum & Praxis, Mainz, Rhineland-Palatinate
  - kfgn Site Operations & Services GmbH (KFGN) - Klinische Forschung Dresden GmbH (KFDD), Dresden, Saxony
  - Herzzentrum Leipzig, Leipzig, Saxony
  - Charite-Universitaetsmedizin Berlin - Campus Benjamin Franklin (CBF), Berlin
  - emovis GmbH, Berlin
  - Gemeinscharftspraxis Dres Jung - Deggingen, Deggingen
  - kfgn Site Operations & Services GmbH (KFGN) - Klinische Forschung Karlsruhe GmbH (KFKA), Karlsruhe
  - Universitaetsklinikum Leipzig - Klinik und Poliklinik fuer Pneumologie, Leipzig
  - KfH Kuratorium fuer Dialyse und Nierentransplantation e.V. - KfH-Nierenzentrum Klaus-Ketzler-Zentrum, Wiesbaden
- Italy (15):
  - Gruppo Humanitas - Humanitas Research Hospital (Istituto Clinico Humanitas), Rozzano, Milan
  - Azienda Ospedaliero-Universitaria Sant'Andrea Roma, Centro Ipertensione, UOC di Cardiologia, Roma, Rome
  - Istituto Nazionale di Riposo e Cura per Anziani (INRCA), Ancona
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna
  - Universita degli Studi Di Brescia - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliero-Universitaria di Ferrara - Arcispedale Sant'Anna, Ferrara
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Azienda Sanitaria Locale 1 (ASL 1) - Ospedale Regionale San Salvatore, L’Aquila
  - Universita degli Studi di Messina - Azienda Ospedaliera Universitaria Policlinico "Gaetano Martino" - Messina, Messina
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - AOU Policlinico di Modena - UO Cardiologia, Modena
  - Azienda Ospedaliera Universitaria (AOU) di Napoli, Napoli
  - Fondazione IRCCS Policlinico San Matteo, - SC Ematologia, Dipartimento Oncoematologico, Pavia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - IRCCS San Raffaele, Rome
- Netherlands (4):
  - Radboud Universiteit - Radboud Universitair Medisch Centrum (Radboudumc), Nijmegen, Gelderland
  - Amsterdam UMC - Locatie AMC (Academisch Medisch Centrum), Amsterdam, North Holland
  - Albert Schweitzer Ziekenhuis - Sliedrecht, Dordrecht, South Holland
  - Universitair Medisch Centrum (UMC) Utrecht - Locatie AZU, Utrecht
- Poland (9):
  - Diamond Clinic Specjalistyczne Poradnie Lekarskie, Krakow, Lesser Poland Voivodeship
  - Velocity Lublin, Lubin, Polska
  - Velocity Skierniewice Sp. z o.o, Skierniewice, Polska
  - ETG Network - Warszawa (European Trial Group), Warsaw, Polska
  - Etyka OÅ>rodek BadaÅ" Klinicznych, Olsztyn, Warmian-Masurian Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny im. Andrzeja Mieleckiego Slaskiego Uniwersytetu Medycznego w Katowicach, Katowice
  - Silmedic Sp. z o.o, Katowice
  - FutureMeds Sp. z o.o. FutureMeds Lodz, Lodz
  - FutureMeds Sp. z o.o. Futuremeds Olsztyn, Olsztyn
- Latin Clinical Trial Center Inc. (LCTC), San Juan, Puerto Rico
- Romania (10):
  - Spitalul Clinic Judetean de Urgenta Tg. Mures, Târgu Mureş, Mureș County
  - Centrul Medicali's Timisoara, Timișoara, Timiș County
  - Centrul Medical Unirea SRL Brasov (Regina Maria), Brasov
  - Delta Health Care SRL Bucuresti - Spitalul Academic Ponderas (Regina Maria), Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Angiocare S.R.L. (Spitalul Ares Cluj-Napoca), Cluj-Napoca
  - Spitalul Clinic Municipal Filantropia Craiova, Craiova
  - Spitalul Clinic Judetean de Urgenta Bihor, Oradea
  - S.C Materna Care SRL Timisoara (Regina Maria), Timișoara
  - Spitalul Clinic Judetean de Urgenta "Pius Branzeu" Timisoara, Timișoara
- Spain (8):
  - Complejo Hospitalario Universitario de Badajoz (CHUB) (Hospital Infanta Cristina), Badajoz
  - Hospital del Mar - Institut Hospital del Mar d'Investigacions Mediques (IMIM), Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Virgen de las Nieves (HUVN), Granada
  - Hospital Clínico San Carlos, Madrid
  - Universidad Autonoma de Madrid (UAM) - Facultad de Medicina - Hospital Universitario Fundacion Jimenez Diaz (UAM-FJD) - Instituto de Investigacion Sanitaria (IIS), Madrid
  - Complejo Hospitalario Universitario de Santiago de Compostela (CHUS) - Hospital Clinico Universitario (University Clinical Hospital), Santiago de Compostela
  - Instituto de Investigacion Sanitaria (INCLIVA), Valencia
- United Kingdom (14):
  - Fowey River Practice - Fowey Surgery, Fowey, Great Britain
  - Queen Mary University of London (QMUL) - Barts and The London School of Medicine and Dentistry - William Harvey Research Institute (WHRI) - William Harvey Heart Centre (WHHC), London, Great Britain
  - Knowle House Surgery, Plymouth, Great Britain
  - The Rame Group Practice (Dr. DAVIS & Partners) - Penntorr Health, Torpoint, Great Britain
  - Cambridge University Hospitals NHS Foundation Trust - Addenbrooke's Hospital (AH), Canterbury, Kent
  - Aberdeen Royal Infirmary, Aberdeen
  - University Hospitals Birmingham NHS Foundation Trust - Birmingham Regional Severe Asthma Service (BRSAS), Birmingham
  - East Kent Hospitals University NHS Foundation Trust, Canterbury
  - Epsom and St Helier University Hospitals NHS Trust, Carshalton
  - Rowden Surgery Rowden Medical Partnership, Chippenham
  - NHS Greater Glasgow and Clyde (NHSGGC), Glasgow
  - Newquay Health Centre, Newquay
  - Sheffield Teaching Hospitals NHS Foundation Trust - Northern General Hospital, Sheffield
  - FutureMeds - Stockton-on-Tees, Stockton-on-Tees

REFERENCES:
- [Derived] Saxena M, Laffin L, Borghi C, Fernandez Fernandez B, Ghali JK, Kopjar B, Polu K, Roger SD, Slingsby BT, Strutz F, Vogt L, Weir MR, Rodman D; Launch-HTN Investigators. Lorundrostat in Participants With Uncontrolled Hypertension and Treatment-Resistant Hypertension: The Launch-HTN Randomized Clinical Trial. JAMA. 2025 Aug 5;334(5):409-418. doi: 10.1001/jama.2025.9413. PMID 40587141